CLINICAL TRIAL: NCT02937896
Title: Comparison of Intranasal Desmopressin vs IV Ketorolac in Renal Colic Patients
Brief Title: Intranasal Desmopressin vs IV Ketorolac in Renal Colic Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kambiz Nasiri, Emergency Medicine Resident, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 688
Record Dates: First submitted 2016-10-12; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Deamino Arginine Vasopressin; Ketorolac; Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketorolac (Experimental): 30mg ketorolac administrated intravenous and 4 puffs nasal Normal Saline.
  Interventions: Drug: Ketorolac; Drug: Normal Saline
- Desmopressin (Active Comparator): 40 microgram nasal desmopressin administrated and 1cc Normal Saline intravenous
  Interventions: Drug: Desmopressin; Drug: Normal Saline

INTERVENTIONS:
Drug: Desmopressin — 40 micrograms Nasal Desmopressin.
  Other Names: Ddavp
  Arms: Desmopressin
Drug: Ketorolac — 30mg intravenous Ketorolac.
  Other Names: Toradol
  Arms: Ketorolac
Drug: Normal Saline — 1cc intravenous Normal Saline.
  Other Names: NaCl
  Arms: Desmopressin
Drug: Normal Saline — 4 puffs nasal Normal Saline.
  Other Names: NaCl
  Arms: Ketorolac

SUMMARY:
The aim of this study is the comparison of efficacy of intravenous ketorolac and intranasal desmopressin in renal colic patients pain control.

DETAILED DESCRIPTION:
40 renal colic patients have been divided into 2 groups randomly, one group has been received 30mg intravenous Ketorolac and 4 puffs nasal Normal Saline while other has been received 40 micrograms nasal Desmopressin and 1cc intravenous Normal Saline. Pain Score before drug administration,also 10, 30 and 60 minutes after drug administration has been measured bye Visual Analogue Scale ( VAS ).

ELIGIBILITY:
Inclusion Criteria:

* renal colic patients

Exclusion Criteria:

* history of hypertension and cardiac disease
* pregnant patients
* use of analgesic within 4 hours before intervention

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pain score | Pain score change from baseline pain score before intervention 10, 30 and 60 minutes after intervention

IPD SHARING:
Plan to Share IPD: Undecided